CLINICAL TRIAL: NCT05281172
Title: Prevention of Alcohol Abuse in Educational Settings (PRVENALC)
Brief Title: Guided Self-Change Prevention Program for Alcohol Abuse in Adolescents in Educational Settings
Acronym: PREVENALC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, Jose Luis Carballo Crespo, PhD, Associate Professor and Researcher, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PID2019-110400RB-I00
Record Dates: First submitted 2022-02-10; First posted 2022-03-16 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Abuse or Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Self-Change therapy (Experimental)
  Interventions: Behavioral: Guided Self-Change therapy (GSC)
- Psychoeducation program about healthy habits (Active Comparator)
  Interventions: Behavioral: Psychoeducation program about healthy habits

INTERVENTIONS:
Behavioral: Guided Self-Change therapy (GSC) — The GSC program follows a motivational cognitive-behavioral approach designed to minimize resistance in drug behavior changes, prevent relapse risk, and increase motivation to quit. The GSC consists of 5 weekly sessions of 50 minutes delivered in groups of 20-25 people.
  Arms: Guided Self-Change therapy
Behavioral: Psychoeducation program about healthy habits — The psychoeducational program will include talks about healthy habits such as physical activity, relaxation, and sleep hygiene. This intervention consists of 5 weekly sessions of 50 minutes delivered in groups of 20-25 people.
  Arms: Psychoeducation program about healthy habits

SUMMARY:
This study corresponds to a pretest-posttest randomized experimental design with two arms. Arm 1 includes Guided Self-Change program, and Arm 2 a psychoeducational program to promote healthy habits. This study aims to analyze the efficacy of a selective and indicated prevention program based on the Guided Self-Change model (GSC) in adolescent alcohol users between 16-18 years. Researchers hypothesize that implementation of GSC therapy will lead to a greater reduction of alcohol drinkers compare with the control condition, and will prevent alcohol abuse after 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 16-18 years old.
* Having inform consent from parents
* Report using alcohol at least once a month during the previous last three months

Exclusion Criteria:

* Participants will be excluded if they refer being diagnosed with a severe mental disorder.
* Have a severe medical illness that will limit participation
* Being under treatment for a psychological of psychiatric problem.
* Meet DSM criteria for Drug dependence to illegal drugs.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 800 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Alcohol use change | Change from baseline up to 5 weeks and two follow-ups at 6 and 12 months post intervention
  Alcohol use will be assessed using the Timeline Follow-Back (Sobell & Sobell, 1992)
Alcohol abuse | Change from baseline to week 5, and at 6 and 12 months post intervention.
  Alcohol abuse will be assessed using the Rutgers Alcohol Problem Index (White & Labouvie, 1989). The global score ranges from 0 to 69, where higher scores represent greater level of alcohol-related problems.
Alcohol dependence | Change from baseline to week 5, and at 6 and 12 months post intervention.
  Alcohol dependence will be assessed with the Alcohol Use Disorder and Associated Disabilities Interview Schedule-5 (Grant et al., 2015).

SECONDARY OUTCOMES:
Drug use | Change from baseline to week 5, and at 6 and 12 months post intervention.
  Assessed with the Drug History Questionnaire (Sobell et al., 1995).
Impulsiveness | Change from baseline to week 5, and at 6 and 12 months post intervention.
  Impulsiveness will be assessed with the Impulsive Behavior Scale (Cyders et al., 2014). The global score ranges from 20 to 80, where higher scores represent greater level of impulsivity.
Sleep quality | Change from baseline to week 5, and at 6 and 12 months post intervention.
  Sleep will be assessed with different sleep measures, such as the Brief version of the Pittsburgh Sleep Quality Index (Sancho-Domingo et al., 2021). The global score of the B-PSQI ranges from 0 to 15, where higher scores represent poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Carballo, PhD, Principal Investigator — Miguel Hernández University of Elche
Locations (1):
- José Luis Carballo, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No